CLINICAL TRIAL: NCT00040872
Title: N8: Dose-Intensive Chemotherapy Plus Biologics in the Treatment of Neuroblastoma
Brief Title: Multiple Therapies in Treating Patients With Advanced Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 00-065; P30CA008748 (NIH); MSKCC-00065; NCI-G02-2083
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Neuroblastoma
Keywords: regional neuroblastoma; disseminated neuroblastoma; recurrent neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; humanized 3F8 anti-GD2 monoclonal antibody; sargramostim; Carboplatin; Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; Isotretinoin; Thiotepa; Topotecan; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: monoclonal antibody 3F8
Biological: sargramostim
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: isotretinoin
Drug: thiotepa
Drug: topotecan hydrochloride
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: conventional surgery
Procedure: drug resistance inhibition treatment
Procedure: peripheral blood stem cell transplantation
Procedure: syngeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Radiation therapy uses high-energy x-rays to damage tumor cells. Biological therapies use different ways to stimulate the immune system and stop cancer cell from growing. Combining different types of therapies may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy, monoclonal antibody therapy, surgery, peripheral stem cell transplantation, radiation therapy, and biological therapy in treating patients who have advanced neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether treatment with multimodality therapy comprising dose-intensive induction chemotherapy, monoclonal antibody 3F8, surgery, myeloablative chemotherapy, autologous or syngeneic bone marrow or peripheral blood stem cell transplantation, radiotherapy, and isotretinoin improves the cure rate in patients with advanced neuroblastoma.
* Determine whether the 2-year progression-free survival (PFS) rate improves to 70% in patients with newly diagnosed advanced neuroblastoma treated with this regimen.
* Determine whether the 2-year PFS rate improves to 40% in patients with previously treated advanced neuroblastoma treated with this regimen.
* Determine the biologic and clinical prognostic factors of neuroblastoma that may guide future research of treatment approaches for this malignancy.

OUTLINE: Patients are stratified according to the following:

* Stratum 1: Patients with previously untreated stage IV disease who are over age 1 at diagnosis, with or without N-myc amplification
* Stratum 2: Patients with previously treated stage IV disease who are over age 1 at diagnosis; or patients with previously treated high-risk disease (e.g., N-myc amplified stage III or IV disease, under age 1 at diagnosis, and with or without prior treatment)
* Intensive induction therapy (courses 1-5): During courses 1, 2, and 4, patients receive cyclophosphamide IV over 6 hours on days 1 and 2 and doxorubicin and vincristine IV continuously on days 1-3. Courses repeat every 21 days. During courses 3 and 5, patients receive etoposide (VP-16) IV over 2 hours on days 1-3 and cisplatin IV over 1 hour on days 1-4. Courses repeat every 35 days. Before proceeding to myeloablative therapy/transplantation, patients in stratum 2 must have received a minimum of 2 courses of chemotherapy if they achieved a complete response (CR) or very good partial response (VGPR) or patients must have received a minimum of 3 courses of chemotherapy if they achieved less than a CR or VGPR.

Patients undergo tumor resection either at diagnosis or after completion of a minimum of 3 courses of chemotherapy (approximately day 63).

Treatment with monoclonal antibody 3F8 (MOAB 3F8) starts after completion of course 3 of intensive induction chemotherapy, preferably after surgical resection or debulking of the primary tumor. Patients receive MOAB 3F8 IV over 90 minutes on days 1-5 of courses 3-5 and on days 1-5 immediately prior to transplantation.

* Harvest: Autologous or syngeneic bone marrow or peripheral blood stem cells (PBSC) are harvested. Patients undergoing PBSC collection receive filgrastim (G-CSF) beginning 2-3 days prior to collection and continuing through the end of collection. For patients without bone marrow involvement at diagnosis, autologous bone marrow or PBSC are harvested after completion of 1-2 courses of induction therapy. For patients with bone marrow involvement at diagnosis, bone marrow or PBSC are harvested after completion of 4 courses of induction therapy, surgery, and completion of 1 course of MOAB 3F8, if bone marrow is in remission. If a patient's bone marrow/PBSC cannot be collected or harvested after completion of induction therapy because of hypoplasia or persistent tumor, bone marrow/PBSC collected or harvested before starting protocol or syngeneic bone marrow/PBSC may be used. If neither of these options is available, patients who do not clear marrow by course 5 have the option of proceeding directly to the posttransplantation therapy phase below, while delaying transplantation until bone marrow is clear.
* Myeloablative therapy/transplantation: Patients receive thiotepa IV over 3 hours on days -8 to -6, topotecan IV over 30 minutes on days -8 to -4, and carboplatin IV over 4 hours on days -5 to -3. Patients undergo autologous or syngeneic bone marrow transplantation (BMT) or PBSC transplantation (PBSCT) on day 0.
* Posttransplantation therapy: Beginning 33 days after BMT/PBSCT, patients receive sargramostim (GM-CSF) subcutaneously on days 1-15 and MOAB 3F8 IV within 90 minutes (beginning approximately 1 hour after initiation of GM-CSF infusion) on days 6-15. Treatment repeats every 28 days for 2 courses.

Beginning 47 days after BMT/PBSCT (on day 14 of course 1 of MOAB 3F8 and GM-CSF), patients receive localized external beam radiotherapy twice daily for 7 consecutive weekdays.

Beginning 82 days after BMT/PBSCT, patients receive alternating courses of oral VP-16 and MOAB 3F8 for a total of 8 courses (total of 4 courses of each drug). Patients receive oral VP-16 3 times daily on days 1-21, with courses repeating every 28 days. Patients receive MOAB 3F8 IV within 90 minutes on days 1-5, with courses repeating every 35 days.

Beginning 222 days after BMT/PBSCT (2-3 weeks after completion of course 4 of oral VP-16), patients receive oral isotretinoin twice daily on days 1-14. Treatment repeats every 28 days for 6 courses.

Beginning on day 243 after BMT/PBSCT, patients receive MOAB 3F8 IV within 90 minutes on days 1-5. Treatment repeats every 28 days for 6 courses.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 49 patients (34 for stratum 1 and 15 for stratum 2) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma by 1 of the following:

  * Histologic confirmation, including immunohistochemical, ultrastructural, or cytogenetic studies
  * Elevated urinary catecholamines plus tumor cells/clumps in the bone marrow
* Poor-risk disease, defined by 1 of the following:

  * Stage IV disease
  * Unresectable primary disease plus N-myc amplification
  * Infant (under age 1) with stage IV disease plus N-myc amplification
* Previously treated disease allowed

PATIENT CHARACTERISTICS:

Age:

* 50 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior allergy to mouse proteins
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior murine antibodies allowed if human anti-mouse antibody (HAMA) titer is less than 1,000 ELISA units/mL

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-06; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Kong V. Cheung, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States